CLINICAL TRIAL: NCT04746131
Title: Safety and Pharmacokinetic Study of IMM0306 in Patients With Refractory or Relapsed CD20-positive B-cell Non-Hodgkin's Lymphoma (B-NHL)
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to the product development strategy change, without any safety concerns, we (the sponsor of the trial) have decided to request to place the IND (#151570) on inactive status.
Sponsor: ImmuneOnco Biopharmaceuticals (Shanghai) Inc. (Other)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMM0306
Record Dates: First submitted 2021-02-04; First posted 2021-02-09 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-04

CONDITIONS: B-cell Non-Hodgkin's Lymphoma
Keywords: IMM0306
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IMM0306 (Experimental): IMM0306 Dose escalation: 0.1mg/kg, 0.2mg/kg, 0.4mg/kg, 0.8mg/kg,1.2mg/kg and 1.6mg/kg through intravenous administration weekly up to 52 weeks.
  Interventions: Drug: IMM0306

INTERVENTIONS:
Drug: IMM0306 — IMM0306 is an bi-specific antibody

SUMMARY:
The purpose of this study is to assess the safety and efficacy of IMM0306-02 in patients with refractory or relapsed CD20-positive B-cell Non-Hodgkin's Lymphoma (B-NHL).

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old
* Diagnosed with B-NHL
* Relapsed after or be refractory to at least 2 line of standard therapy

Exclusion Criteria:

* Active central nervous system (CNS) metastases
* Positive Direct Antiglobulin Test (DAT)
* Active autoimmune disorder
* Skin disorders that do not requires hormone replacement therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2024-04-11 (Estimated); Study Completion 2024-04-11 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of IMM0306 as measured by incidence of DLTs (Dose Limiting Toxicity) | End of Study (52 Weeks)
  DLT is defined as one of the following toxicities occurring during the DLT assessment for Cycle 1.

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Huang, MD, Study Director — VP，Clinical Development
Locations (1):
- The Christ Hospital, Cincinnati, Ohio, United States